CLINICAL TRIAL: NCT02394366
Title: Effects of Topical Herbal Salve on Cutaneous Oxygenation and Peripheral Blood Flow
Brief Title: Topical Salve for Skin Oxygenation and Blood Flow
Acronym: OHS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Ryan Bradley, Associate Professor, National University of Natural Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 01202015
Record Dates: First submitted 2015-03-13; First posted 2015-03-20 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Skin Oxygenation; Peripheral Perfusion
Keywords: Skin oxygenation; peripheral perfusion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Original Healing Salve (Puremedy, Inc.) including 1x homeopathic dilutions of Calendula, Echinacea, and Sambucus extracts, plus extracts from pine and Balsam fir; acute effects only
  Interventions: Other: Original Healing Salve (OHS)
- Control (Placebo Comparator): Original Health Salve olive oil and beeswax base only without homeopathic or herbal extracts; acute effects only
  Interventions: Other: OHS base only

INTERVENTIONS:
Other: Original Healing Salve (OHS) — Topical salve (Puremedy, Inc.)
  Arms: Active
Other: OHS base only — Olive and beeswax salve base
  Arms: Control

SUMMARY:
Delayed wound healing leads to increased risk for infection, and thus increased risk for morbidity and mortality. Skin oxygen delivery and peripheral blood flow predict wound healing. The investigators will conduct a double-masked, placebo-controlled cross-over clinical pilot trial in order to evaluate the effects of a topical, homeopathic/herbal salve (Original Healing Salve, Puremedy, Inc.) on skin oxygenation and peripheral blood flow.

DETAILED DESCRIPTION:
Delayed wound healing leads to increased risk for infection, and thus increased risk for morbidity and mortality. Skin oxygen delivery and peripheral blood flow predict wound healing. In order to evaluate the effects of a topical, homeopathic/herbal salve (Original Healing Salve, Puremedy, Inc.) on skin oxygenation and peripheral blood flow, the investigators will conduct a double-masked, placebo-controlled cross-over clinical pilot trial with randomized testing order to evaluate the effects of the salve on cutaneous oxygen saturation (TcPO2) and ankle-to-brachial pressure index (ABPI). The investigators will recruit thirty-two participants in two cohorts to participate, one with and one without type 2 diabetes, who are otherwise generally healthy without active wounds, ulcers or skin rashes. Both TcPO2 and ABPI will be measured before and after the application of both the homeopathic/herbal salve ("active"), and before and after the application of the inert salve base ("placebo"). Analyses will compare pre/post changes in TcPO2 and ABPI before and after application of the active salve within the same visit, and also compare the changes from the active salve to the before and after changes in TcPO2 and ABPI measured from the placebo salve. If the Original Healing Salve improves cutaneous oxygenation and/or ABPI, future research may evaluate the formula specifically for wound healing and antimicrobial effects. Thus the proposed research is a pilot study targeting mechanistic outcomes, which predict potential clinical efficacy. The proposed research is significant, as lower cost, more effective treatments are needed to improve wound healing and reduce the morbidity associated with the complications of delayed wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes without known complications, i.e., eye damage (retinopathy), nerve damage (diabetic peripheral neuropathy), kidney damage (diabetic kidney disease), or heart damage (recent myocardial infarction or severe congestive heart failure)
* Age ≥ 18 and ≤ 75
* Willing and able to give informed consent
* Able to follow protocol and attend visits
* Able to read and write English

Exclusion Criteria:

* Active malignancy, excluding basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ of the cervix. If present, dermal cancers may not be located on or around the testing sites.
* A recent cardiovascular event (e.g., myocardial infarction, stroke ≤ six months prior to screening visit), current coronary artery disease, angina, stage III or IV congestive heart failure, or stated history of coronary bypass surgery or heart stent placement.
* Current active diabetic ulcers.
* History of diabetic neuropathy.
* Diagnosis of type 2 diabetes for longer than 10 years.
* Diagnosis of type 1 diabetes.
* Established diagnosis of peripheral artery disease (PAD) or intermittent claudication.
* Established diagnosis of peripheral venous disease (PVD) or chronic venous insufficiency.
* Active rash, wound, or ulcer on lower leg, including psoriasis or eczema.
* Presence of edema > +1; pitting or non pitting.
* Currently taking any of the following beta-blocker medications (due to potential impact on peripheral vasodilation): acebutolol (Sectral®), atenolol (Tenormin®), betaxolol (Kerlone®), bisoprolol fumarate (Zebeta®, Ziac®), carvedilol (Coreg®),metoprolol (Lopressor®, Toprol XL®), nadolol (Corgard®), nebivolol (Bystolic®), penbutolol (Levatol®), propranolol (Hemangeol®, Inderal LA® Inderal XL®, InnoPran XL®), esmolol (Brevibloc), sotalol (Betapace, Sorine), labetalol (Normodyne, Trandate), pindolol (Visken).
* Currently taking any of the following cholinergic medications (due to potential impact on peripheral vasodilation): acetylcholine, atropine, bethanechol (Urecholine®), donepezil (Aricept®), ipratropium bromide (Atrovent®), neostigmine (Prostigmine®), nicotine (Nicoderm®, Nicotrol®), oxybutynin (Ditropan®), physostigmine, pilocarpine (Salagen®), pralidoxime (Protopam®), succinylcholine (Anectine®), tiotropium bromide (Spiriva®, Tiova®), tolterodine (Detrol®), vecuronium (Norcuron®).
* Allergy to any ingredient found in the study products: pine resin, balsam fir resin, elder (Sambucus) flower and bark, marigold (Calendula), cone flower (Echinacea), olive oil, safflower oil or beeswax.
* Walking Impairment Questionnaire Speed Scores between 0-18 due to risk for PAD (21).
* Walking Impairment Questionnaire Distance Scores between 0-19 due to risk for PAD (21).
* Presence of an unstable and/or significant medical disorder that would compromise the participant's safety to take part in the trial.
* Use of tobacco products, e-cigarettes, nicotine patches and/or nicotine gum
* Scleroderma
* Raynaud's
* Planned elective surgery within the next 6 weeks
* Pregnant, nursing, or planning a pregnancy within the next 6 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Transcutaneous oxygen pressure (TcPO2) | 30 minutes
  Change in TcPO2 will be compared between 0 min and 30 mins between Active and Placebo arms

SECONDARY OUTCOMES:
Ankle-to-Brachial Pressure Index (ABPI) | 30 minutes
  Change in ABPI will be compared between 0 min and 30 mins between Active and Placebo arms

OTHER OUTCOMES:
Trend in TcPO2 | 0 to 30 minutes
  Longitudinal trend in TcPO2 will be evaluated via measurements taken at 5 minutes intervals over 30 minutes

REFERENCES:
- [Background] Browne AC, Sibbald RG. The diabetic neuropathic ulcer: an overview. Ostomy Wound Manage. 1999 Jan;45(1A Suppl):6S-20S; quiz 21S-22S. PMID 10085972
- [Background] Cina C, Katsamouris A, Megerman J, Brewster DC, Strayhorn EC, Robison JG, Abbott WM. Utility of transcutaneous oxygen tension measurements in peripheral arterial occlusive disease. J Vasc Surg. 1984 Mar;1(2):362-71. doi: 10.1067/mva.1984.avs0010362. PMID 6481885
- [Background] Blake DF, Young DA, Brown LH. Transcutaneous oximetry: normal values for the lower limb. Diving Hyperb Med. 2014 Sep;44(3):146-53. PMID 25311321 (Retraction: PMID 27044466 Diving Hyperb Med. 2016 Mar;46(1):54)
- [Background] Andrews KL, Dib MY, Shives TC, Hoskin TL, Liedl DA, Boon AJ. Noninvasive arterial studies including transcutaneous oxygen pressure measurements with the limbs elevated or dependent to predict healing after partial foot amputation. Am J Phys Med Rehabil. 2013 May;92(5):385-92. doi: 10.1097/PHM.0b013e3182876a06. PMID 23478457
- [Background] Reddy KK, Grossman L, Rogers GS. Common complementary and alternative therapies with potential use in dermatologic surgery: risks and benefits. J Am Acad Dermatol. 2013 Apr;68(4):e127-e135. doi: 10.1016/j.jaad.2011.06.030. Epub 2011 Sep 3. PMID 21890235
- [Background] Umscheid CA, Mitchell MD, Doshi JA, Agarwal R, Williams K, Brennan PJ. Estimating the proportion of healthcare-associated infections that are reasonably preventable and the related mortality and costs. Infect Control Hosp Epidemiol. 2011 Feb;32(2):101-14. doi: 10.1086/657912. PMID 21460463
- [Background] Cesarone MR, Belcaro G, Rohdewald P, Pellegrini L, Ledda A, Vinciguerra G, Ricci A, Ippolito E, Fano F, Dugall M, Cacchio M, Di Renzo A, Hosoi M, Stuard S, Corsi M. Improvement of signs and symptoms of chronic venous insufficiency and microangiopathy with Pycnogenol: a prospective, controlled study. Phytomedicine. 2010 Sep;17(11):835-9. doi: 10.1016/j.phymed.2010.04.009. Epub 2010 Jun 25. PMID 20579863
- [Background] Fife CE, Smart DR, Sheffield PJ, Hopf HW, Hawkins G, Clarke D. Transcutaneous oximetry in clinical practice: consensus statements from an expert panel based on evidence. Undersea Hyperb Med. 2009 Jan-Feb;36(1):43-53. PMID 19341127
- [Background] Aboyans V, Ho E, Denenberg JO, Ho LA, Natarajan L, Criqui MH. The association between elevated ankle systolic pressures and peripheral occlusive arterial disease in diabetic and nondiabetic subjects. J Vasc Surg. 2008 Nov;48(5):1197-203. doi: 10.1016/j.jvs.2008.06.005. Epub 2008 Aug 9. PMID 18692981
- [Background] Mathieu D, Mani R. A review of the clinical significance of tissue hypoxia measurements in lower extremity wound management. Int J Low Extrem Wounds. 2007 Dec;6(4):273-83. doi: 10.1177/1534734607310299. PMID 18048873
- [Background] Humphreys ML, Stewart AH, Gohel MS, Taylor M, Whyman MR, Poskitt KR. Management of mixed arterial and venous leg ulcers. Br J Surg. 2007 Sep;94(9):1104-7. doi: 10.1002/bjs.5757. PMID 17497654
- [Background] Belcaro G, Cesarone MR, Errichi BM, Ledda A, Di Renzo A, Stuard S, Dugall M, Pellegrini L, Gizzi G, Rohdewald P, Ippolito E, Ricci A, Cacchio M, Cipollone G, Ruffini I, Fano F, Hosoi M. Diabetic ulcers: microcirculatory improvement and faster healing with pycnogenol. Clin Appl Thromb Hemost. 2006 Jul;12(3):318-23. doi: 10.1177/1076029606290133. PMID 16959685
- [Background] Duran V, Matic M, Jovanovc M, Mimica N, Gajinov Z, Poljacki M, Boza P. Results of the clinical examination of an ointment with marigold (Calendula officinalis) extract in the treatment of venous leg ulcers. Int J Tissue React. 2005;27(3):101-6. PMID 16372475
- [Background] Khmel'nitskii OK, Simbirtsev AS, Konusova VG, McHedlidze GSh, Fidarov EZ, Paramonov BA, Chebotarev VY. Pine resin and Biopin ointment: effects on cell composition and histochemical changes in wounds. Bull Exp Biol Med. 2002 Jun;133(6):583-5. doi: 10.1023/a:1020290010605. PMID 12447472
- [Background] McDermott MM, Liu K, Guralnik JM, Martin GJ, Criqui MH, Greenland P. Measurement of walking endurance and walking velocity with questionnaire: validation of the walking impairment questionnaire in men and women with peripheral arterial disease. J Vasc Surg. 1998 Dec;28(6):1072-81. doi: 10.1016/s0741-5214(98)70034-5. PMID 9845659
- [Background] Conlon KC, Sclafani L, DiResta GR, Brennan MF. Comparison of transcutaneous oximetry and laser Doppler flowmetry as noninvasive predictors of wound healing after excision of extremity soft-tissue sarcomas. Surgery. 1994 Mar;115(3):335-40. PMID 8128357
- [Background] White RA, Nolan L, Harley D, Long J, Klein S, Tremper K, Nelson R, Tabrisky J, Shoemaker W. Noninvasive evaluation of peripheral vascular disease using transcutaneous oxygen tension. Am J Surg. 1982 Jul;144(1):68-75. doi: 10.1016/0002-9610(82)90604-3. PMID 7091534
- [Background] Ratliff DA, Clyne CA, Chant AD, Webster JH. Prediction of amputation wound healing: the role of transcutaneous pO2 assessment. Br J Surg. 1984 Mar;71(3):219-22. doi: 10.1002/bjs.1800710320. PMID 6697129
- [Background] Karanfilian RG, Lynch TG, Zirul VT, Padberg FT, Jamil Z, Hobson RW 2nd. The value of laser Doppler velocimetry and transcutaneous oxygen tension determination in predicting healing of ischemic forefoot ulcerations and amputations in diabetic and nondiabetic patients. J Vasc Surg. 1986 Nov;4(5):511-6. PMID 2945936
- [Background] Kram HB, Appel PL, Shoemaker WC. Multisensor transcutaneous oximetric mapping to predict below-knee amputation wound healing: use of a critical Po2. J Vasc Surg. 1989 Jun;9(6):796-800. doi: 10.1067/mva.1989.vs0090796. PMID 2657122